CLINICAL TRIAL: NCT02384889
Title: Targeting Polyamines Using DFMO in Persons With Type 1 Diabetes: A Randomized, Double-Masked, Placebo-Controlled Phase I Study to Evaluate the Safety, Tolerability, and Initial Pharmacodynamics of Multiple Ascending Doses
Brief Title: DFMO in Children With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Linda DiMeglio, MD, Professor, Indiana University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1411735324
Record Dates: First submitted 2015-02-12; First posted 2015-03-10 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Eflornithine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Difluoromethylornithine (Experimental): Subjects may be given daily dose of DFMO
  Interventions: Drug: Difluoromethylornithine
- Placebo (Placebo Comparator): Subjects may be given daily dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Difluoromethylornithine — Active Therapy with DFMO
  Other Names: DFMO
  Arms: Difluoromethylornithine
Drug: Placebo — Placebo Comparitor
  Other Names: Comparitor
  Arms: Placebo

SUMMARY:
This study is a multicenter, double-blind, placebo-controlled, 2:1 randomly assigned, phase 1 clinical trial for individuals with type 1 diabetes. It is a blinded dose-ranging study enrolling patients with new onset type 1 diabetes with documented continued residual C-peptide production. After a 4 week screening and run-in period during which eligibility will be determined and glycemic control optimized, subjects will have a 3-month double-masked treatment period with either DFMO or placebo. After a 3 month wash-out period the durability of effect will be assessed. Subjects will be randomly assigned (6 to DFMO; 3 to placebo in each cohort) to 1 of 4 sequential dose cohorts.

DETAILED DESCRIPTION:
This study is repurposing alpha difluoromethylornithine (DFMO) in order to characterize its effects in persons with new onset type 1 diabetes. In preliminary studies in mice, inhibition of polyamine synthesis with DFMO preserved β-cell insulin production and delayed diabetes onset. Polyamine modulation has the potential to improve β cell health in persons with T1D. The investigators propose that decreasing polyamine synthesis in persons with new onset T1D will improve markers of ß cell health and function.

This double-masked, placebo-controlled dose-finding randomized multiple ascending dose study will include a 1-month screening period; a 3-month double-masked treatment period; and a 3-month follow-up period. Subjects will be randomly assigned to 1 of 4 sequential dose cohorts: DFMO at nominal (starting) doses of 125 mg/m2 per day, 250 mg/m2 per day, 500 mg/m2 per day, and then 750 mg/m2 per day. Dose escalation will be done based upon whether any dose limiting toxicities are observed and whether any suggestion of effect on biomarkers of β-cell stress is observed. At a maximum dose, the cohort will be expanded in order to estimate biomarker activity. If there is no suggestion of effect and no dose-limiting toxicity 750 mg/m2 per day, a 750 mg per day group will be enrolled. Regardless of the dose we expand, the investigators will evaluate efficacy of treatment on the primary and secondary outcomes. The primary outcome endpoint in this study will be the safety of the doses. In particular, the dose-limiting toxicities known to be potential side effects of DFMO (thrombocytopenia, neutropenia, anemia, audiometric impairment) will be reviewed and monitored by an internal safety review committee before each cohort is enrolled. Secondary outcomes will include biomarkers of beta cell stress, measures of insulin production/glycemia. Exploratory outcomes will include flow cytometry assessment of B- and T-cell subsets, quantification of polyamine intake and excretion, and pharmacokinetic DFMO concentrations. Completion of this study will facilitate future work in studies of DFMO or other inhibitors of pathways that influence intracellular polyamine levels, including non-steroidal inflammatory agents, and novel polyamine transport inhibitors. .

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 12-40 years of age with a clinical diagnosis of T1D within 2 - 8 months after diagnosis at the time of visit 2.
2. Random non-fasting C-peptide level of >0.2 pmol/mL at visit 1.
3. Positive for any one of the following diabetes-related autoantibodies (mIAA, GADA, IA-2A, or ZnT8A)
4. Treatment naïve of any immunomodulatory agent
5. Normal hearing at screening, defined as acceptable results of pure-tone audiometry (<20 decibel [dB] baseline thresholds for frequencies 250, 500, 1000, and 2000 Hz

Exclusion Criteria:

1. Presence of severe, active disease that interferes with dietary intake or requires the use of chronic medication, with the exception of well-controlled hypothyroidism and mild asthma not requiring oral steroids. Presence of any psychiatric disorder that will affect ability to participate in study.
2. Diabetes other than T1D
3. Chronic illness known to affect glucose metabolism (e.g. Cushing syndrome, polycystic ovarian disorder, cystic fibrosis) or taking medications that affect glucose metabolism (e.g. steroids, metformin)
4. Inability to swallow pills
5. Psychiatric impairment or current use of anti-psychotic medication
6. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results.
7. Hematologic abnormalities at screening (anemia, leukopenia (particularly neutropenia), or thrombocytopenia)
8. Impaired renal function (assessed by history and BUN/Creatinine, DFMO is renally excreted)
9. Female participants of child-bearing age must not be pregnant and agree to use an effective form of birth control or be abstinent during the study period.
10. BMI >95% for age and sex

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2015-04; Primary Completion 2019-10-07 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities | 6 month
  Low platelet counts, low white blood cell counts, low hemoglobin, severe abdominal pain/diarrhea, hearing loss

OTHER OUTCOMES:
Changes in Serum Markers of Beta Cell Stress | 6 months
  Observed Changes in pro-insulin and c-peptide measured from blood

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Riley Hospital for Children, Indianapolis, Indiana
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Children's Hospital of Wisconsin, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Sims EK, Kulkarni A, Hull A, Woerner SE, Cabrera S, Mastrandrea LD, Hammoud B, Sarkar S, Nakayasu ES, Mastracci TL, Perkins SM, Ouyang F, Webb-Robertson BJ, Enriquez JR, Tersey SA, Evans-Molina C, Long SA, Blanchfield L, Gerner EW, Mirmira RG, DiMeglio LA. Inhibition of polyamine biosynthesis preserves beta cell function in type 1 diabetes. Cell Rep Med. 2023 Nov 21;4(11):101261. doi: 10.1016/j.xcrm.2023.101261. Epub 2023 Nov 1. PMID 37918404
- [Derived] Robertson MA, Padgett LR, Fine JA, Chopra G, Mastracci TL. Targeting polyamine biosynthesis to stimulate beta cell regeneration in zebrafish. Islets. 2020 Sep 2;12(5):99-107. doi: 10.1080/19382014.2020.1791530. Epub 2020 Jul 25. PMID 32715853